CLINICAL TRIAL: NCT04448938
Title: RESting-state Functional MRI in Patients With Optic Neuritis for ANticipation of reCovEry
Acronym: RESONANCE
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 2020-A01560-39
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Neuritis
MeSH Terms: conditions — Neuritis | interventions — Visual Acuity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- optic neuritis
  Interventions: Other: MRI; Other: visual acuity
- control
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — The MRI examination will be performed on a 3T multi-parametric MRI. Compared to the standard protocol, patients will benefit from an additional sequence of f-mRI, called resting state, and performed before injection of gadolinium contrast agent.
  A consultation with an ophthalmologist will also be carried out the same day, at the Adolphe de Rothschild Foundation.
  The subjects of the control group who agreed to participate will benefit from an MRI examination which will include, in addition to the sequences planned for these patients according to their indications, the two non-injected sequences which will be performed on patients with suspected NO.
Other: visual acuity — Patients with NO will be seen in consultation by an ophthalmologist during a follow-up visit approximately 6 months after diagnosis. During this consultation, an OCT, a visual field and the measurement of visual acuity will be performed. This visit and the examinations carried out correspond to the usual care of patients suffering from NO and followed at the Adolphe de Rothschild Foundation Hospital
  Groups: optic neuritis

SUMMARY:
When patients arrive in the waiting room of the MRI department, patients will be given the briefing note explaining the purpose of the study and how it is going. During the consultation, the radiologist will check the inclusion and non-inclusion criteria, and will take the time to answer all of the patient's questions about the study. If the patient agrees to participate in the research, the investigating doctor will obtain his consent.

The MRI examination will be performed on a 3T multi-parametric MRI. Compared to the standard protocol, patients will benefit from an additional sequence of f-mRI, called resting state, and performed before injection of gadolinium contrast agent.

A consultation with an ophthalmologist will also be carried out the same day, at the Adolphe de Rothschild Foundation. During this visit, an OCT examination (optical coherence tomography), a visual field as well as the measurement of visual acuity will be carried out, in accordance with the treatment usually practiced at the Adolphe de Rothschild Foundation.

The subjects of the control group who agreed to participate will benefit from an MRI examination which will include, in addition to the sequences planned for these patients according to their indications, the two non-injected sequences which will be performed on patients with suspected NO.

The possible existence of visual problems in the subjects of the control group will also be asked to them by interrogation. No eye exams or follow-up visits are planned, and control group participation will end after the MRI scan.

Patients with NO will be seen in consultation by an ophthalmologist during a follow-up visit approximately 6 months after diagnosis. During this consultation, an OCT, a visual field and the measurement of visual acuity will be performed. This visit and the examinations carried out correspond to the usual care of patients suffering from NO and followed at the Adolphe de Rothschild Foundation Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Clinical suspicion of optic neuritis
* Benefiting from an MRI for exploration of optic neuritis
* Affiliate or beneficiary of a social security scheme
* Having received informed information about the study and having given their express consent to participate in the study

Exclusion Criteria:

* Contraindication to absolute or relative MRI (in particular, pregnant or breastfeeding women)
* History of amblyopia
* Any pre-existing pathology leading to a decrease in vision (e.g. retinitis pigmentosa, AMD, etc.)
* Patient benefiting from a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical suspicion of NO who must perform an MRI for the diagnosis of NO. A control group will also be set up to compare the visual functional networks of patients with NO with those of a sample of subjects free from NO.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The ophthalmological functional recovery will be assessed by measuring the low contrast visual acuity on the Early Treatment Diabetic Retinopathy study scale (ETDRS scale). | 6 months
  ETDRS charts presents a serie of 70 letters. The visual acuity letter score is equal to the total number of letters read correctly at 4.0 m. The score ranged to 20/10 (best visual acuity) to 20/20 000 (worst visual acuity).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation A De Rothschild, Paris, PARIS, France

IPD SHARING:
Plan to Share IPD: No